CLINICAL TRIAL: NCT00072605
Title: VRC 204 A Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of a Multiple Strain Ebola DNA Plasmid Vaccine, VRC-EBODNA012-00-VP, in Adult Volunteers
Brief Title: Experimental Ebola Vaccine Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040028; 04-I-0028
Record Dates: First submitted 2003-11-04; First posted 2003-11-05 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2007-08-22

CONDITIONS: Hemorrhagic Fever, Ebola; Healthy
Keywords: Healthy; T Cells; Immunity; Hemorrhagic Fever; Healthy Volunteer; HV
MeSH Terms: conditions — Hemorrhagic Fever, Ebola; Hemorrhagic Fevers, Viral

INTERVENTIONS:
Drug: VRC-EBODNA012-00-VP

SUMMARY:
This study will test the safety of an experimental vaccine developed to protect against Ebola virus infection and to determine if the vaccine induces an immune response to the virus. The Ebola virus causes a disease called Ebola hemorrhagic fever. Symptoms begin with fever and muscle aches and progress to breathing problems, severe bleeding, kidney problems, and shock. The infection may be mild, but it can also lead to death. The vaccine used in this study is made from small parts of Ebola genetic material. It cannot cause Ebola hemorrhagic fever to develop in those who receive it.

Healthy volunteers 18 to 44 years of age may be eligible for this study. Candidates will be screened with a medical history, physical examination, and laboratory tests, and complete an "assessment of understanding" questionnaire to show that they understand the study.

Depending on their order of entry into the study, participants are assigned to receive one of three vaccine doses or placebo. The first group receives the lowest dose (2 milligram) of vaccine or placebo. If this dose is safe, then the second group receives 4 mg, and if this dose is safe, the third group receives 8 mg. Injections are given in a muscle in the upper arm. Participants receive three injections, each 4 weeks apart (on study days 0, 28, and 56).

Participants record their temperature and symptoms in a diary card for 7 days following each injection. They return to the clinic 2 to 3 days after each injection and then 2 weeks after each injection until study week 10. Additional follow-up visits are then scheduled at weeks 12, 24, 38, and 52. At each visit, participants provide a blood and urine sample for testing and have their vital signs, and lymph nodes checked, their weight measured, and their symptoms reviewed. Additional laboratory tests may be requested between visits.

DETAILED DESCRIPTION:
This is a Phase I, randomized, placebo-controlled, dose-escalation study of an Ebola DNA plasmid vaccine. The hypothesis is that the vaccine will be safe for human administration and elicit immune responses to Ebola. Primary objectives are to evaluate the safety and tolerability of the investigational vaccine and the secondary objective is to evaluate immune responses. Randomization assignment will be blinded to subjects, clinical investigators and laboratory investigators.

ELIGIBILITY:
* INCLUSION CRITERIA:

A volunteer must meet all of the following inclusion criteria:

1. 18 to 44 years old.
2. Available for follow-up for the duration of the study (12 months).
3. Able to provide proof of identity to the acceptance of the study clinician completing the enrollment process.
4. Completion of an Assessment of Understanding prior to enrollment and verbalize understanding of all questions answered incorrectly.
5. Able and willing to complete the informed consent process.
6. Willing to receive HIV test results and willing to abide by NIH guidelines for partner notification of positive HIV results.
7. Willing to donate blood for sample storage.
8. In good general health without clinically significant medical history.
9. Physical examination and laboratory results without clinically significant findings within the 28 days prior to enrollment.

   Laboratory Criteria within 28 days prior to enrollment:
10. Hematocrit equal to 34% for women; 38% for men.
11. Normal fibrinogen levels, D-dimer immunoassay less than 2.0 microg/mL, and RBC morphology without evidence of microangiopathic hemolysis.
12. WBC count: Non-African Americans: equal to 3,300-12,000 cells/mm3, African-Americans: equal to 2,500 - 12,000 cells/mm3 (in the absence of clinical or pathological etiology).
13. Differential either within institutional normal range or accompanied by site physician approval.
14. Total lymphocyte count: Non-African Americans: equal to 800 cells/mm3, African Americans: equal to 650 cells/mm3 (in the absence of clinical or pathological etiology)
15. Platelets within institutional normal limits.
16. Prothrombin time and activated partial thromboplastin time (PT, PTT) within institutional normal range.
17. Alanine aminotransferase (ALT) (also called SGPT) = upper limit of normal range
18. Serum creatinine = upper limit of normal range
19. Negative Food and Drug Administration (FDA)-approved HIV blood test
20. Negative hepatitis B surface antigen (HbsAg)
21. Negative antibody to hepatitis C virus (anti-HCV), or negative HCV PCR if the anti-HCV is positive.
22. Normal urinalysis defined as negative glucose, negative or trace protein, and negative hemoglobin by dipstick.

    Female-Specific Criteria:
23. Negative pregnancy test (urine or serum) for women presumed to be of reproductive potential.
24. A female participant must meet one of the following criteria:

No reproductive potential because of menopause (one year without menses) or because of a hysterectomy, bilateral oophorectomy, or tubal ligation,

or

Participant agrees to be heterosexually inactive at least 21 days prior to enrollment and throughout the duration of the study,

or

Participant agrees to consistently practice contraception at least 21 days prior to enrollment and throughout the duration of the study by one of the following methods:

* condoms, male or female, with or without a spermicide
* diaphragm or cervical cap with spermicide
* intrauterine device
* contraceptive pills or patch, Norplant, Depo-Provera or other FDA-approved contraceptive method
* male partner has previously undergone a vasectomy for which there is documentation

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following conditions apply.

Women:

1. Breast-feeding.

   Volunteer has received any of the following substances:
2. Immunosuppressive or cytotoxic medications within the past six months with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis
3. Blood products within 120 days prior to HIV screening.
4. Immunoglobulin within 60 days prior to HIV screening.
5. Live attenuated vaccines within 30 days prior to initial study injection.
6. Investigational research agents within 30 days prior to initial study injection.
7. Medically indicated subunit or killed vaccines, e.g. influenza, pneumococcal, or allergy treatment with antigen injections, within 14 days prior to initial study injection.
8. Current anti-TB prophylaxis or therapy.

   Volunteer has a history of any of the following clinically significant conditions:
9. Serious adverse reactions to vaccines, such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain.
10. Autoimmune disease or immunodeficiency.
11. Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or intravenous corticosteroids.
12. Diabetes mellitus (type I or II), with the exception of gestational diabetes.
13. Thyroid disease including history of thyroidectomy and diagnoses that required medication within the past 12 months.
14. Serious angioedema episodes within the previous 3 years or requiring medication in the previous two years.
15. Hypertension that is not well controlled by medication or is more than 145/95 at enrollment.
16. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
17. Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study.
18. Seizure disorder other than: 1) febrile seizures under the age of two, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) a singular seizure not requiring treatment within the last 3 years.
19. Asplenia or any condition resulting in the absence or removal of the spleen.
20. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder requiring therapy that has not been well controlled by medication for the past two years; disorder requiring lithium; or suicidal ideation occurring within five years prior to enrollment
21. Any medical, psychiatric, or social condition, or occupational or other responsibility that, in the judgment of the investigator, would interfere with or serve as a contraindication to protocol adherence or a volunteer's ability to give informed consent.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27
Dates: Start 2003-10-30; Study Completion 2007-08-22

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Birmingham K, Cooney S. Ebola: small, but real progress. Nat Med. 2002 Apr;8(4):313. doi: 10.1038/nm0402-313. No abstract available. PMID 11927920